CLINICAL TRIAL: NCT05868447
Title: Investigation of the Relationship Between Perioperative Blood Transfusion and Intraoperatively Monitored Oxygen Reserve Index (ORI) in Patients Scheduled for Vertebral Stabilization Surgery
Brief Title: Relationship Between ORI and Blood Transfusion in Spinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Asiye Demirel, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011- KAEK- 25 2022/12-10
Record Dates: First submitted 2023-05-08; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Hemorrhage
Keywords: Oxygen reserve index; Blood transfusion; vertebrae stabilization surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Stabilization surgery — hourly blood gas analysis and hemoglobin and hematocrit control and blood transfusion will be performed when necessary
  If a low pO2 value is observed in the blood gas, the fi02 values or fresh gas flow will be increased.

SUMMARY:
Concerns about the necessity and risks of blood transfusions have led to the search for new noninvasive monitoring methods. Oxygen reserve index (ORI), one of them, is a dimensionless index ranging from 0.00 (no reserve) to 1.00 (maximum reserve) according to oxygenation reserve status, and it is also a non-invasive and continuous measurement parameter. Some studies have examined ORi as an indicator for early detection of hypoxemia. There are reports in the literature that ORi and Pa02 values measured noninvasively during surgery are early precursors for desaturation and hypoxia.Researces aimed to investigate the relationship between perioperative blood transfusions and ORI in vertebral stabilization surgeries performed by the same surgical team in our clinic.

DETAILED DESCRIPTION:
With the increase in the elderly population in the world, the incidence of vertebral deformities is increasing and vertebral surgery has become one of the most commonly performed surgeries. Blood loss in vertebral and spinal canal deformity surgeries varies according to the surgical procedure, duration of operation and type of anesthesia. With the increase in blood loss, blood and blood product transfusion also increases. Although many technical and pharmacological methods have been applied to reduce blood transfusion in surgical patients, there is still no consensus on when to transfuse, and there are still institutional and individual differences in transfusion practices. In the literature, there are studies showing that some centers never use blood for the same surgery in patients, while in other centers blood is almost always used [4]. This has led to the comment that "Blood transfusion is a practice that takes place according to the physician, not the patient." The World Health Organization (WHO) defines anemia as hemoglobin (Hb) concentration <13 g/dl for men and <12 g/dl for women. Although these Hb concentrations stated in the literature try to define the lowest acceptable hemoglobin, transfusion practices are based on multiple physiologic parameters (tachycardia, hypotension, ST segment changes) rather than an isolated laboratory measurement (Hb and hematocrit values), The decision to transfuse blood is known to be difficult to standardize as it has to be made taking into account the need for increased oxygen extraction rate, new-onset wall motion abnormalities on transesophageal echocardiography, cardiac output and oxygen content of arterial blood, central venous oxygen saturation, base deficit, lactate level, etc.). The decision to transfuse blood is based on the hope of increasing tissue oxygen delivery (DO2), followed by cellular oxygenation. Improving DO2 has been shown to reduce both morbidity and mortality in the perioperative period. Tailoring DO2 to O2 consumption using specific targets seems promising. The common criterion used to start blood transfusion therapy is to determine the Hb level and to show that the DO2 has fallen to the critical Hb level, which is assumed to be compromised. With this view triggered by the Hb level detected at the critical level, transfusion is performed and it is seen that the Hb level is increased to a safe level after transfusion. Although it can be easily demonstrated that transfusion therapy increases Hb level and consequently DO2, it requires further research to determine how this treatment reflects on the general oxygen supply/consumption balance. Indeed, for this purpose, monitoring of mixed central venous oxygen saturation (SvO2) is a prerequisite. This method, which requires a pulmonary artery catheter, is currently used in very limited situations and indications and central venous saturation (ScvO2) value is generally used instead of SvO2.

Anesthesia management of the patients included in the study and the interventional procedures to be performed will be decided by the responsible anesthesiologist.

The initial ORI value of the patient will be determined as PO2 value between 100-120 mmHg in arterial blood gas (ABG) and will be recorded on the case report form every 15 minutes. The preoperative Hb value will also be recorded on the case report form, and in patients with intraoperative expected blood loss >500 ml and for whom blood transfusion is foreseen, the hemoglobin value and ORI value will be recorded by the responsible anesthesiologist at the time of the indication of erythrocyte transfusion. Accordingly, the relationship between the initial ORI value and the ORI value at the time of the decision for erythrocyte transfusion will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age in ASA I-III risk class
* Patients who will undergo vertebral stabilization surgery at 3 levels or more under general anesthesia (lumbar disc herniation, lumbar spinal stenosis, lumbar spondylolisthesis and other lumbar spine pathologies)
* who are expected to lose >500 ml of blood
* Patients who require arterial catheter placement for continuous monitoring of blood pressure and/or analysis of arterial blood gas during surgery

Exclusion Criteria:

* Patients with coagulation disorders, thrombocytopenia, liver and kidney disease
* Patients receiving regular anticoagulant and antiplatelet therapy
* Patients who will undergo revision surgery
* Patients who will undergo surgery due to spinal tumor or infection
* Patients with perioperative tranexamic acid and/or antifibrinolytic use
* Patients with preoperative hemoglobin values <12 g/dl in women and <13 g/dl in men or patients with preoperative anemia due to hemoglobinopathies (e.g. thalassemia, sickle cell disease anemia)
* Patients with congestive heart failure
* Inability to attach the sensor due to deformity of the fingers
* Inability to attach the sensor due to hypoperfusion of the fingers: thalassemia, sickle cell disease anemia)
* Patients with congestive heart failure
* Inability to wear the sensor due to deformity of the fingers
* Patients who would show an inadequate signal due to hypoperfusion of the fingers were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elective patients planned stabilization surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative ORI values | Perioperative process (2-5 hours)
  Monitoring ORI values at the beginning of surgery and values measured every 15 minutes during surgery

SECONDARY OUTCOMES:
Perioperative blood transfusion prediction | Perioperative process (2-5 hours)
  To measure the ORI values from the beginning of the case until the end of the case with a finger probe from the patient's finger with the Oxygen reserve index (ORI) monitoring device in patients who will undergo vertebral stabilization surgery and to determine how much the ORI value decreases compared to the beginning of surgery when the patient bleeds and to answer the question of whether the decrease can predict the erythrocyte transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Asiye A Demirel, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No